CLINICAL TRIAL: NCT06600230
Title: The Effect of Pelvic Floor-Based Training on Young Women With Dysmenorrhea
Brief Title: Effect of Pelvic Floor-Based Training on Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, tuba kolaylı, Lecturer, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61351342/2023-41
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dysmenorrhea
Keywords: dysmenorrhea; pelvic floor; physiotherapy; exercise education
MeSH Terms: conditions — Dysmenorrhea | interventions — Educational Status; Exercise; Hot Temperature

STUDY DESIGN:
Intervention Model Description: Before - after trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Pelvic floor and exercise training was given by physiotherapists.
  Interventions: Other: Education and exercise
- Control group (Active Comparator): Classical self-methods such as hot application were applied
  Interventions: Other: Self-method like resting or heat

INTERVENTIONS:
Other: Education and exercise — Training including information on pelvic floor and dysmenorrhea and exercise practices were given both theoretically and practically by physiotherapists.
  Arms: Interventional group
Other: Self-method like resting or heat — Classical self-methods such as rest and heat application were applied.
  Arms: Control group

SUMMARY:
The aim of this study is to examine the effect of patient education, knowledge levels and dysmenorrhea symptoms in young women with primary dysmenorrhea. The main question it aims to answer is the questions are as follows:

1. Is patient education effective in improving symptoms in young women with primary dysmenorrhea?
2. Is there a relationship between knowledge level and symptoms in young women with primary dysmenorrhea?

Participants will:

After the training group was given the training in 2 sessions, the participants were asked to apply the exercises in which the training was given. The control group applied conventional self-methods when dysmenorrhea symptoms occurred. The evaluations were made before the training and at the end of the first menstrual cycle.

DETAILED DESCRIPTION:
Dysmenorrhea is pain that occurs during menstruation due to cramps in the uterus. It is one of the most common causes of pelvic pain, especially experienced by young women. primary dysmenorrhea is distinguished from secondary dysmenorrhea by the occurrence of pain in women with normal pelvic anatomy without any pathology or physiological etiology. In the management of primary dysmenorrhea, non-pharmacological treatment methods such as lifestyle changes, sleep and nutrition changes, exercise, and physiotherapy applications are used in addition to pharmacological treatments. The aim of this study is to examine the effect of patient education on the pelvic floor knowledge levels and dysmenorrhea symptoms in young women with primary dysmenorrhea. In this study, participants were divided into two groups: the education group and the control group. The evaluations were made before the education and after the first menstrual cycle. The "Statistical Package for Social Sciences (SPSS) Statistics 23.0 (SPSS Inc, Chicago, USA) program will be used in the analysis of the study data. The change in numerical variables over time in the treatment and control groups and the group-time interaction will be examined with "two-way repeated measures variance analysis". The "Chi-Square Test" will be used to examine the relationship between categorical variables. The relationship between numerical variables will be examined with the "Spearman rho correlation coefficient". The probability of error will be accepted as (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with primary dysmenorrhea
* Being between the ages of 18-35
* Having a regular menstrual cycle
* Volunteering to participate in the study

Exclusion Criteria:

* Not having a history of endometriosis or gynecological pathology •
* Having a history of gynecological disease or surgery
* Having a neurological or musculoskeletal problem

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 month
  VAS , is used to determine the subjective perceived pain intensity. People with pain are expected to mark the pain intensity they feel on a 0-10 cm scale. The value of '0' indicates no pain, while the value of '10' indicates the most severe pain. VAS is used to assess menstrual pain intensity in individuals with primary dysmenorrhea.
Pelvic Floor Health Knowledge Test | 1 month
  PFHKT, was developed in Turkish by Wala'a and Çelenay to measure the knowledge level of people about the pelvic floor. Each correct answer to the questions in the test is given '1' point, each wrong or blank answer is given '0' point. The lowest score that can be obtained from the scale is '0' and the highest score is '29'. An increase in the score obtained in the test, which has been studied for validity and reliability, indicates a higher level of knowledge.

SECONDARY OUTCOMES:
Dysmenorrhea Affect Scale | 1 month
  DAS, was developed to provide a holistic assessment of dysmenorrhea. The scale includes health perception/management, nutrition and metabolism, excretion, activity and exercise, sleep and rest, cognition and perception, self-perception, role and relationship, sexuality and productivity in Gordon's functional health patterns model. There are items based on the topics of coping with stress and stress tolerance, values and beliefs. As the participants' scores on the scale increase, their level of being affected by dysmenorrhea also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No